CLINICAL TRIAL: NCT07177352
Title: Master Screening Study to Determine Individuals With Potential Trial Eligibility for Alzheimer's Disease Studies as Assessed by Biomarker Status and Cognition
Brief Title: Screening Study to Determine Individuals With Potential Trial Eligibility for Alzheimer's Disease Studies
Acronym: TRAVELLER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WP45722
Record Dates: First submitted 2025-09-15; First posted 2025-09-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Alzheimers Disease
Keywords: Early Alzheimers Disease; Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Arm (Other): Participants will be assessed for their concentration of pTau217 in blood and cognitive score in the International Shopping List Test (ISLT).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants will have their blood drawn and cognitive score measured by the ISLT.

SUMMARY:
This study is a pre-screening process used to assess participants' potential eligibility for Roche interventional Alzheimer's disease studies.

ELIGIBILITY:
Inclusion Criteria:

- Report of objective or subjective memory concerns (by the participant and/or their informant) within the last year with or without a previous clinical diagnosis of MCI or dementia due to AD.

Exclusion Criteria:

* Dependency in basic activities of daily living (bADLs) due to cognitive impairment
* Visual or auditory impairment that would prevent them from performing the cognitive assessments (eyeglasses and hearing aids are permitted)
* Any self-reported evidence or known diagnosis of a neurological or neurodegenerative condition that may lead to cognitive impairment other than AD
* History of severe, clinically significant central nervous system trauma
* Any serious medical condition that precludes a participant's safe participation and completion of a clinical study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13000 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2035-07-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of pTau217 in Blood on Day1 | Day 1
Cognitive score in ISLT on Day 1 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (202):
- United States (66):
  - Banner Alzheimer?s Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Sun Valley Research Center, Inc., Imperial, California
  - Inglewood Clinicals, Inglewood, California
  - Irvine Center for Clinical Research, Irvine, California
  - Healthy Brain Clinic, Long Beach, California
  - Oakland Clinical, Oakland, California
  - Riverside Clinical, Riverside, California
  - Syrentis Clinical Research, Santa Ana, California
  - Cenexel California Neuroscience Research, LLC, Sherman Oaks, California
  - Yale University, New Haven, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - K2 Medical Research-Winter Garden, Clermont, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Visionary Investigators Network- Neurology Aventura, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park/Orlando, Orlando, Florida
  - Conquest Research - Lake Nona, Orlando, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Axiom Brain Health LLC, Tampa, Florida
  - Charter Research - Lady Lake/The Villages, The Villages, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Alzheimer's Research and Treatment Center - Columbus, Columbus, Georgia
  - Accel Research Sites-NeuroStudies, Decatur, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - RE:Cognition (Chicago), Chicago, Illinois
  - Great Lakes Clinical Trials Chicago d/b/a Flourish Research Andersonville, Chicago, Illinois
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Adams Clinical Boston, Boston, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Adams Clinical Watertown, Watertown, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Washington University School of MedicineClinical Translational Research Unit, St Louis, Missouri
  - The Cognitive and Research Center of New Jersey, Ridgewood, New Jersey
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - IMA Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Basil Clinical, Laurelton, New York
  - Weill Cornell Medical College, New York, New York
  - Adams Clinical Harlem, New York, New York
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - Adams Clinical Bronx, The Bronx, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - Ohio State University, Columbus, Ohio
  - Summit Research Network Inc., Portland, Oregon
  - Flourish Research ? Philadelphia, Plymouth Meeting, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Palmetto Clinical Trials, Summerville, South Carolina
  - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - K2 Medical Research - Nashville, Nashville, Tennessee
  - Gadolin Research, LLC, Beaumont, Texas
  - South Texas Research Institute - Brownsville, Brownsville, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Kerwin Research Center, LLC, Dallas, Texas
  - South Texas Research Institute - Edinburg, Edinburg, Texas
  - Re:Cognition Health - Fort Worth, Fort Worth, Texas
  - Re:Cognition Health - Houston, Houston, Texas
  - Mt.Olympus Medical Research, Katy, Texas
  - El Faro Health and Therapeutics, Rio Grande City, Texas
  - Sana Research, LLC, Arlington, Virginia
  - Re:Cognition Health, Fairfax, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
- Argentina (4):
  - INECO Neurociencias Orono, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundacion Scherbovsky, Mendoza
  - Sanatorio del Sur S.A., San Miguel de Tucumán
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - KaRa Institute of Neurological Diseases, Macquarie Park, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Heidelberg Repatriation Hospital, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Brazil (5):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Clinica Clinilive ltda, Maringá, Paraná
  - Instituto do Cerebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica, Joinville, Santa Catarina
  - Centro de Pesquisas Clinicas - CPCLIN, São Paulo, São Paulo
- Canada (15):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Richmond Clinical Trials, Richmond, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - Parkwood Institute, Mental Health Care Building, London, Ontario
  - Bruyère Health Research Institute, Ottawa, Ontario
  - The Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Centricity East York, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Clinique Memoire de Montreal, Montreal, Quebec
  - Genge Partners Inc., Montreal, Quebec
  - Alpha Recherche Clinique, Québec
- China (16):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital - Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - The second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Nanjing Brain Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
- Italy (10):
  - A. O. U. Federico II, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione Santa Lucia IRCCS, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ospedale Isola Tiberina - Gemelli Isola, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - AOU Policlinico Giaccone, Palermo, Sicily
  - AO di Perugia - Ospedale S. Maria della Misericordia, Perugia, Umbria
- Japan (20):
  - Brain Attack Center Ota Memorial Hospital, Hiroshima
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Kobe University Hospital, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Kochi Medical School Hospital, Kochi
  - National Hospital Organization Utano National Hospital, Kyoto
  - Mishuku Hospital, Meguro-Ku
  - Mie University Hospital, Mie
  - Okayama City Hospital, Okayama
  - Rijikai Medical Corporation Katayama Medical Clinic, Okayama
  - Kotobuki Social Medical Corporation Tominaga Clinic, Osaka
  - Memory Clinic Ochanomizu, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Higashi-Shinjuku Clinic, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tokyo
  - P-One Clinic, Tokyo
  - Yamagata Tokusyukai Hospital, Yamagata
- Poland (21):
  - ProNeuro Centrum Medyczne, ?ory
  - Uniwersytet Medyczny w Lodzi, ?ód?
  - Syberka-ClinHouse Sp. z o.o., B?dzin
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - Centrum Medyczne Neuromed Sp. z.o.o., Bydgoszcz
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gda?sk
  - Uniwersyteckie Centrum Kliniczne;Klinika Neurologii Doros?ych, Gdansk
  - Neuro-Care Gabriela Klodowska, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Clinical Research Center Sp. z o.o. MEDIC-R Spó?ka Komandytowa, Późna
  - Nmedis sp. z o.o., Rzeszów
  - Centrum Medyczne Medyk, Rzeszów
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - O?rodek Badawczo-Naukowo-Dydaktyczny Chorób Ot?piennych w ?cinawie, Ścinawa
  - Centrum Medyczne NeuroProtect, Warsaw
  - ETG Neuroscience Sp. z o.o., Warsaw
  - Centrum Leczenia Zaburzen Pamieci, Warsaw
  - NZOZ WCA, Wroc?aw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanislawa SzyszkoSUM w Katowicach, Zabrze
- University of Puerto Rico - Medical Science Campus, San Juan, Puerto Rico
- South Korea (11):
  - Chonnam National University Hospital, Gwangju
  - St. Vincent's Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Hanyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
  - Korea University Guro Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Medical Center, Suwon
- Spain (15):
  - Hospital de Dénia;Servicio de Neurología, Denia, Alicante
  - Fundació Hospitalàries Martorell;Neurology, Martorell, Barcelona
  - Hospital Mutua De Terrasa, Terrassa, Barcelona
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Fundación ACE, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Policlínica Guipuzkoa, Donosti-San Sebastián
  - Hospital San Cecilio, Granada
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario la Fe, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Neurology, Kwei Shen
  - Taipei Medical University - Shuang Ho Hospital - Neurology, New Taipei City
  - China Medical University Hospital, North Dist.
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No